CLINICAL TRIAL: NCT05594771
Title: Comparative Study of the Loading Dose Administrated Via Epidural Needle or Epidural Catheter for Labor Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB-20220306-R
Record Dates: First submitted 2022-10-22; First posted 2022-10-26 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2022-10

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- epidural needle (Experimental): the loading dose for labor analgesia administrated via epidural needle before the catheter insertion.
  Interventions: Procedure: epidural needle
- epidural catheter (Active Comparator): the loading dose for labor analgesia administrated via the epidural catheter.
  Interventions: Procedure: epidural catheter

INTERVENTIONS:
Procedure: epidural needle — the loading dose for labor analgesia administrated via epidural needle before the catheter insertion
  Arms: epidural needle
Procedure: epidural catheter — the loading dose for labor analgesia administrated via epidural catheter
  Arms: epidural catheter

SUMMARY:
Epidural anesthesia (EP) is widely used for labor analgesia. Time to onset of adequate pain relief of EP technique for labor analgesia may be 15 to 20 minutes.More rapid injection is often passible through the needle compared to catheter and could enhance the spread of medication within the epidural space.There is lack of research assessing the onset of labor analgesia with a large priming dose of local anesthetic through the epidural needle compared with the epidural catheter.

DETAILED DESCRIPTION:
The epidural analgesia was performed in the left lateral decubitus position at the L3-L4 or L2-L3 interspace using a 18 G Tuohy needle. The epidural space was accessed by the loss of resistance to air or saline (2ml or less) technique.

In the epidural needle group, after identification of epidural space, a dose of 3 ml of 0.1%ropivacaine with 0.3ug/ml sufentanil was given via the epidural needle ,3 minutes later labor analgesia was initiated with 15ml of 0.1 ropivacaine with 0.3ug/ml sufentanil over 30 seconds via the epidural needle, and then the catheter was inserted 3-5cm into the epidural space. In the epidural catheter group, the catheter was inserted 3-5cm into the epidural space after identification of epidural space, a dose of 3 ml of 0.1% ropivacaine with 0.3ug/ml sufentanil was given via the epidural catheter, 3minutes later labor analgesia was initiated with 15ml of 0.1%ropivacaine with 0.3ug/ml sufentanil as the same of group N.

ELIGIBILITY:
Inclusion Criteria:

1. healthy, term (37-42 weeks' gestation),
2. nulliparous women with singleton
3. patients in active labor with a cervical dilation <5cm who planned labor analgesia

Exclusion Criteria:

1. any contraindication to neuraxial anesthesia,
2. body mass index>50kg/m2,
3. VAS <50mm on a 100-mm visual analog pain scales during an active contraction, 4. pregnancy-related diseases (ie, gestational hypertension, gestational diabetes, and preeclampsia),

5. the participants were in the event of an inadvertent dural puncture using the epidural needle, 6.fetal heart abnormity before labor analgesia.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 276 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
The time to onset of labor analgesia | 8 months
  Compare time of onset of labor analgesia and adequate analgesia was defined as VAS score<10mm in the presence of contraction.

SECONDARY OUTCOMES:
VSA scores | 8 months
  the Visual Analog Scale (VAS) on a 100-mm scale is measured during the labor .
number of PCEA bolus requests | 8 months
  the numbers of the patient -controlled epidural anangesia(PCEA) bolus of 5 ml with 15 minute lockout.
analgesia drug ( ropivacaine) requests | 8 months
  The total ropivacaine dose is recorded and is divided by the hours.

CONTACTS AND LOCATIONS:
Overall Officials: Xinzhong Chen, Study Director — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Department of Anesthesiology, Women's Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Chen X, Tang Y, Yu Q, Sun L, Li H, Wang L, Jiao C, Chen X. Comparative study of labour analgesia onset with injection of loading dose through epidural needle versus catheter: A prospective, double-blinded, randomised clinical trial. Eur J Anaesthesiol. 2025 Feb 1;42(2):113-121. doi: 10.1097/EJA.0000000000002077. Epub 2024 Oct 16. PMID 39744745